CLINICAL TRIAL: NCT02630043
Title: A Phase I Trial of Tolcapone Alone and in Combination With Oxaliplatin in Patients With Relapsed or Refractory Neuroblastoma
Brief Title: Trial of Tolcapone With Oxaliplatin for Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of study enrollment
Sponsor: Giselle Sholler (Other)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Study Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMTRC011
Record Dates: First submitted 2015-12-04; First posted 2015-12-15 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Tolcapone; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tolcapone and Oxaliplatin (Experimental): Subjects will receive oral tolcapone at their assigned dose level on each day of this 21-day cycle.
  Oxaliplatin will be given at 100 mg/m2 IV on Day 1 of Cycle 2 through 5 and any subsequent 21-day cycle.
  Interventions: Drug: Tolcapone; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Tolcapone — Tolcapone is an oral agent that will be administered every day of each 21-day cycle during Cycle 1 and in combination with oxaliplatin during cycles 2-5 given IV on Day 1 of each 21-day cycle.
  Other Names: Tasmar
Drug: Oxaliplatin — Oxaliplatin will be given starting in Cycle 2 at 100 mg/m2 IV on Day 1 of each 21-day cycle
  Other Names: Eloxatin

SUMMARY:
The purpose of this research study is to evaluate an investigational drug (Tolcapone) alone and in combination with oxaliplatin, for relapsed and refractory neuroblastoma. Tolcapone is approved by the U.S. Food and Drug Administration (FDA) for adults, but is an investigational drug in this study because it has not been approved in pediatrics for this indication. Oxaliplatin, although a drug approved by the FDA for other cancers, is investigational for treatment of neuroblastoma in this study. This study will look at the safety and tolerability of tolcapone in combination with oxaliplatin as well as the tumors response to this study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≤ 21 years at the time of study entry.
2. Diagnosis: Histologic verification at either the time of original diagnosis or relapse of neuroblastoma.
3. Disease Status: Patients must have ONE of the following:

   * Any episode of recurrent disease following completion of aggressive multi-drug frontline therapy.
   * Any episode of progressive disease during aggressive multi-drug frontline therapy.
   * Primary resistant/refractory disease detected at the conclusion of at least 4 cycles of aggressive multidrug induction chemotherapy on or according to a high-risk neuroblastoma protocols.
4. Measurable or evaluable disease, including at least one of the following: measureable tumor by CT or MRI; a positive MIBG, or PET scan; positive bone marrow biopsy/aspirate.
5. Current disease state must be one for which there is currently no known curative therapy
6. A negative urine or serum pregnancy test is required for female subjects of child bearing potential (onset of menses or ≥13 years of age).
7. Organ Function Requirements:

   * Subjects must have adequate liver function as defined by:

     * AST and ALT ≤ upper limit of normal
     * Serum bilirubin must be ≤ 2.0 mg/dl
   * Subjects must have adequate Bone Marrow function defined as:

For patients without bone marrow involvement:

• Peripheral absolute neutrophil count (ANC) >750/uL

* Subjects must have adequate renal function
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for 90 days after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

* Lansky score <50%
* BSA (m2) of <0.5
* Prior Therapy- Patients must have fully recovered from the acute toxic effects of all prior anti- cancer chemotherapy and be within the following timelines:

  * Myelosuppressive chemotherapy: Must not have received within 2 weeks of enrollment onto this study (6 weeks if prior nitrosourea).
  * Hematopoietic growth factors: At least 5 days since the completion of therapy with a growth factor.
  * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the Study Chair.
  * Immunotherapy: At least 6 weeks since the completion of any type of immunotherapy, e.g. tumor vaccines.
  * Monoclonal antibodies: At least 7 days or 3 half-lives, whichever is longer, must have elapsed since prior treatment with a monoclonal antibody.
  * XRT: At least 14 days since the last treatment except for radiation delivered with palliative intent to a non-target site.
  * Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and ≥ 2 months must have elapsed since transplant.
* Investigational Drugs: Subjects who have received another investigational drug within the last 14 days are excluded from participation.
* Subjects with CNS lesions are excluded
* Subjects with a history of depression, anxiety, or psychotic disorders (due to tolcapone adverse event profile).
* Subjects that are pregnant or breastfeeding an infant.
* Subjects that cannot swallow tablets.
* Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Ages: 0 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
  To determine the safety and tolerability of tolcapone alone and in combination with oxaliplatin at 4 dose levels of tolcapone

SECONDARY OUTCOMES:
Determine the Overall Response Rate (ORR) of Participants using RECIST criteria | 3 years
  To determine the overall response rate (ORR) by the presence of radiologically assessable disease by cross-sectional imaging and in MIBG or PET scans.
Determine the Progression Free Survival (PFS) of Participants using days until progression | 3 years
  To evaluate the activity of tolcapone in combination with oxaliplatin in relapsed or refractory neuroblastoma based on:
  Progression free survival (PFS)
To evaluate the drug levels and pharmacokinetics (PK) of Tolcapone from blood samples at multiple time points within the first 24 hours on study based on Plasma half-life (t1/2). | 24 hours
  Tolcapone plasma concentration-time data will be determined for all subjects enrolled on study.
To evaluate the drug levels and pharmacokinetics (PK) of Tolcapone from blood samples at multiple time points within the first 24 hours on study based on Plasma clearance (Cl). | 24 hours
  Tolcapone plasma concentration-time data will be determined for all subjects enrolled on study.
To evaluate the drug levels and pharmacokinetics (PK) of Tolcapone from blood samples at multiple time points within the first 24 hours on study based on Vd. | 24 hours
  Tolcapone plasma concentration-time data will be determined for all subjects enrolled on study.
To evaluate the drug levels and pharmacokinetics (PK) of Tolcapone from blood samples at multiple time points within the first 24 hours on study based on Peak Plasma Concentration (Cmax) | 24 hours
  Tolcapone plasma concentration-time data will be determined for all subjects enrolled on study.
To evaluate the drug levels and pharmacokinetics (PK) of Tolcapone from blood samples at multiple time points within the first 24 hours on study based on Area Under the Curve (AUC). | 24 hours
  Tolcapone plasma concentration-time data will be determined for all subjects enrolled on study.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Foley, MD, Study Chair — Corewell Health West
Locations (9):
- United States (9):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- See also: Consortium website — http://www.beatcc.org

DOCUMENTS (1):
  • Informed Consent Form (2016-05-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT02630043/ICF_000.pdf